CLINICAL TRIAL: NCT05682001
Title: The Molecular Pathogenesis Study of Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jin Yang, Professor, Eye & ENT Hospital of Fudan University
Other Study IDs: CMP
Record Dates: First submitted 2022-12-06; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Cataract; Pathogenesis
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anterior lens capsule tissues from cataract patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DC group: Anterior lens capsule tissues from DC patients
- ARC group: Anterior lens capsule tissues from ARC patients
- NC group: anterior lens capsules collected from three age-matched transparent crystals of cadaveric eyes

SUMMARY:
To study the molecular pathogenesis of cataract and explore possible treatments，anterior lens capsules were collected from cataract patients

DETAILED DESCRIPTION:
Anterior lens capsules were collected from the patients with DC and ARC, and transparent crystals of cadaveric eyes. M6A epitranscriptomic microarray was performed to investigate the altered m6A modifications and determine the differentially expressed mRNAs. The potential role of dysregulated m6A modification levels was predicted through Gene Ontology and Kyoto Encyclopedia of Genes and Genomes pathway enrichment analyses. Real-time polymerase chain reaction was performed to identify the dysregulated expression of RNA methyltransferases, demethylases, and readers.

ELIGIBILITY:
Inclusion Criteria:

* diabetic cataract
* underwent cataract surgery

Exclusion Criteria:

* Combined with other eye diseases
* underwent other eye surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anterior lens capsule tissues from cataract patients with diabetes mellitus more than 10 years, patients with age related cataract, and transparent crystals of cadaveric eyes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
m6A modification of mRNAs | 1 month
  Epitranscriptomic microarray analysis reveals the differential m6A modification of mRNAs in DC samples
expression level of mRNAs | 1 month
  the m6A microarray analyses provide data for mRNA expression levels
levels of methylated mRNA | 1 month
  in vitro validation of the diverse expression levels of methylated mRNA
levels of RNA methyltransferase | 1 month
  in vitro validation of the diverse expression levels of RNA methyltransferase

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, PhD, Principal Investigator — Eye & ENT Hospital
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No